CLINICAL TRIAL: NCT02307994
Title: Effectiveness and Safety of uFSH for Severe Oligospermia or Azoospermia:A Multi-center,Open,Randomized,Interventional,and Phase4 Trial in China
Brief Title: Clinical Research on Effectiveness and Safety of Treatment of Severe Oligospermia or Azoospermia With uFSH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIVZON-R-14-01
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-08

CONDITIONS: Oligospermia; Azoospermia
Keywords: infertility
MeSH Terms: conditions — Oligospermia; Azoospermia; Infertility

ARMS (1):
- 75IU uFSH (Experimental): 75IU uFSH (Livzon Pharm Group Inc., China) being injected into severe oligospermia patients or azoospermia patients every 3 days for 6 months
  Interventions: Drug: 75IU uFSH

INTERVENTIONS:
Drug: 75IU uFSH

SUMMARY:
The purpose of this study is to determine whether uFSH is effective and safe in the treatment of male patients with severe oligospermia or azoospermia.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 20~35.
* They accorded with diagnostic criteria of severe oligospermia or azoospermia.
* They had'nt been treated with drug which could improve sperm count and quality one month before observation，otherwise,they should have a elution for 1 month before the study.

Exclusion Criteria:

* Gram-positive bacteria ,Chlamydia trachomatis,Ureaplasmaurealyticum,or mycoplasma hominis were detected in their semen.
* Subjects addicted to drug，tobacco，or alcohol.
* Subjects had heat,chemicals,radioactive material,or toxic contact history within a year.
* Subjects were under treatment of gonadotropin,anabolic steroid,chemotherapeutic drugs,or nonsteroidal anti-inflammatory drugs .
* Subjects combined with cardiovascular, liver, kidney ,or hematopoietic system severe primary disease,or mental disease.
* Subjects were allergic or on uFSH allergy,or under the treatment of other drugs for infertility .
* Subjects did not meet the inclusion criteria, did not according to the prescribed medication, were unable to judge the efficacy ,had incomplete information, or affected the efficacy or safety judgment.
* Subjects were IHH patients

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Sperm density | 6 month
(A + B)grade sperm and sperm activity rate | 6 month
A grade sperm | 6 month
semen volume | 6 month
sex hormone levels | 6 month
testis volume | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China